

# **COHORT STUDY PROTOCOL**

An international non-randomized time-bound prospective observational cohort study addressing the epidemiology and management of Small Bowel Obstruction

Study period: November 01st 2023 - May 31st 2024

ClinicalTrials.gov Registration: NCTxxxxxxx

# **Table of contents**

| ESTES SnapSBO Study Steering Committee | 3 |
|-------------------------------------------------------------------|----|
| Introduction | 4 |
| Scope | 5 |
| Key Study Dates | 6 |
| Definitions | 7 |
| Methods | 8 |
| Summary | 8 |
| Primary Objective | 8 |
| Methods for identifying patients | 8 |
| Research Questions | 9 |
| Inclusion and Exclusion Criteria | 10 |
| Center eligibility | 10 |
| Patient follow-up | 10 |
| Data completion | 11 |
| Missing data and retrospective patient entry | 11 |
| Data collection system and information governance | 11 |
| Local approvals | 11 |
| Authorship | 12 |
| Publication of data | 12 |
| Data governance | 12 |
| Financial arrangements | 12 |
| Reference list | 13 |
| REDCap® Data Collection Instruments | 14 |
| Data Collection Instrument 1 - Patient and Centre Demographics | 14 |
| Data Collection Instrument 2 - Patient demographics | 14 |
| Data Collection Instrument 3 - Patient past medical history | 15 |
| Data Collection Instrument 4 - Patient past surgical history | 15 |
| Data Collection Instrument 5 - Patient past SBO history | 16 |
| Data Collection Instrument 6 - Current episode Symptoms and signs | 16 |
| Data Collection Instrument 7 - Initial Complementary Exams | 17 |
| Data Collection Instrument 8 - Current episode, course evolution | 18 |
| Data Collection Instrument 9 - Current episode Surgery | 19 |
| Data Collection Instrument 10 - Current episode, Final outcome | 19 |

# **ESTES SnapSBO Study Steering Committee**

| Name | Country | Center | Email |
|---|---|---|---|
| Isidro Martinez Casas, MD PhD FACS hFEBS(Em Surg) | Spain | Hospital Universitario Virgen del Rocio, Sevilla | isidromartinez@me.com |
| Gary Alan Bass, MD MBA PhD<br>FEBS (Em Surg) | USA /<br>Ireland | University of Pennsylvania, Philadelphia | gary.bass@pennmedicine.upenn.edu |
| Shahin Mohseni, MD PhD FACS<br>hFEBS(Em Surg) | Sweden/ | Orebro University Hospital, Orebro | mohsenishahin@yahoo.com |
| Hayato Kurihara, MD hFEBS(Em<br>Surg) | Italy | Fondazione IRCCS Ca' Granda Ospedale<br>Maggiore Policlinico di Milano | hayato.kurihara@gmail.com |
| Matteo María Cimino, MD | Italy | Fondazione IRCCS Ca' Granda Ospedale<br>Maggiore Policlinico di Milano | Matteo.cimino@policlinico.mil.it |
| Lewis J Kaplan, MD FACS FCCM<br>FCCP | USA | University of Pennsylvania, Philadelphia;<br>Corporal Michael J. Cresencz Veterans Affairs<br>Medical Center, Philadelphia | Lewis.Kaplan@pennmedicine.upenn.edu |

### Introduction

Multi-center, 'snapshot' cohort studies or audits have the ability to gather large patient numbers in short time periods from many hospitals. They allow exploration of differences in patients, techniques and management across the cohort to identify areas of practice variability that may result in apparent differences in outcome. As such, whilst not providing true evidence of efficacy or the impact of a particular variable, they can be hypothesis-generating and can identify areas warranting further study in future randomized controlled trials<sup>1</sup>.

The European Society of Trauma and Emergency Surgery has recognized the strengths of this form of research, as well as its power in bringing together surgeons and emergency surgical units across multiple regions or countries for a common research goal, thus strengthening an active network of research participation across Europe.

## Scope

Small bowel obstruction (SBO) and its complications are frequently seen in patients admitted through the Emergency Departments of all acute care hospitals<sup>2</sup>.

There is variation in the optimal use of imaging, the appropriate timing and duration of non-operative management attempts, anti-microbial therapies and the criteria for surgical management, which results in heterogeneity in approaches and outcomes across international clinical centers. The expected number of SBO cases in most clinical centers is predictable, enabling a suitable sized cohort of patients to be gathered in the snapshot audit.

This 'ESTES snapshot audit' -a prospective observational cohort study- has a dual purpose. Firstly, as an epidemiological study, it aims to uncover the burden of disease. Secondly, it aims to demonstrate current strategies employed to diagnose and treat these patients. These twin aims will serve to provide a 'snapshot' of what we are doing now, but will also be hypothesis-generating while providing a rich source of patient-level data to allow further analysis of particular clinical question.

# **Key Study Dates**

| 06 may 2023 | Snapshot Launch at ECTES 2023, Ljubljana. Center enrolment and local IRB submission |
|---|---|
| 01 november 2023<br>- 01 may 2024 | Patient enrolment. Ninety (90) consecutive day enrollment within this six (6) month window |
| 01 may 2024 | Final day for new patient enrolment |
| 31 July 2024 | Final day of patient follow-up (60 days from admission on 01 may 2024) |
| 01 August 2024 -<br>01 September 2024 | Local data validation, completion, and final upload |
| 01 september 2024 | REDCap® database locked; this is the deadline for data submission and center inclusion. |





### **Definitions**

**Mechanical small bowel obstruction (SBO):** An intrinsic, extrinsic or endoluminal process which narrows or occludes the bowel lumen and delays the passage of luminal contents.

**Ileus:** Functional motility disorder characterized by adynamic paralytic bowel, leading to many of the same symptoms of mechanical obstruction, but without a single site of obstruction demonstrable on imaging. Common causes include recent abdominal surgery, medications such as opiates, and electrolyte disturbances<sup>2</sup>.

**Complete SBO:** Obstruction with no passage of luminal contents beyond the point of obstruction<sup>3</sup> (Appendix A).

**Partial SBO:** Incomplete obstruction with luminal narrowing but some contents continue to pass through the intestine. This is distinguished from complete obstruction by the continued passage of bowel movements and flatus, and a non-peritonitic abdominal exam<sup>3</sup>.

**Small bowel dilatation:** Luminal diameter of >3 cm.

**Transition zone:** Short segment area between dilated proximal bowel and decompressed distal bowel. Sometimes called a transition point and is radiographic evidence of SBO.

**Bowel compromise:** when there is ischemia or injury that has led to necrosis and/or perforation of the bowel wall<sup>4</sup>.

**Adhesions:** Fibrous tissue that connects surfaces or organs within the peritoneal cavity that are normally separated. Such adhesions are the results of an adaptive healing response of the peritoneum upon tissue handling or contact with blood or purulence, but also caused by other conditions like radiotherapy, endometriosis, inflammation or local response to tumors<sup>5</sup>.

**Virgin abdomen:** abdomen of a patient without prior surgery. Although there is no consensus in the literature about radiotherapy, known peritoneal inflammatory disease or primary abdominal wall hernias, in our study we will consider only those non-operated inside the definition<sup>6</sup>.

Water Soluble Oral Contrast (WSOC) challenge: a combined diagnostic study and therapeutic intervention utilized in the evaluation and management of small bowel obstruction.

### **Methods**

#### Summary

Prospective audit of consecutive patients admitted in Emergency Department for mechanical small bowel obstruction over a 3 month period. The audit shall include unscheduled patient admissions from November 2023 until May 2024 as outlined in 'Key Study Dates'.

As this is an observational cohort audit, no change to normal patient management is required.

#### **Primary Objective**

To explore differences in patients, management and outcomes across the entire cohort to identify areas of practice variability resulting in apparent differences in outcome warranting further study. The outcomes that the study will examine are:

- Incidence of small bowel obstruction by etiology.
- Differences in clinical presentation.
- Diagnostic work-up.
- Non-operative management strategies.
- Time to surgery and outcomes.
- Complications related to disease and/or therapies within 60 post-operative days.
- Length of Emergency Department and Hospital stay.
- Re-admission within 6 months for related conditions.

#### Methods for identifying patients

Multiple methods may be used according to local circumstances/staffing:

- 1. Daily review of emergency department (non-operative) and operating room lists.
- 2. Daily review of team handover sheets / emergency admission lists / ward lists.
- 3. Review of operating room logbooks.
- 4. Use of electronic systems to flag any readmissions of patients identified and treated.

#### Research Questions

#### **Primary Research Questions**

- What is the global incidence of SBO?
- What are the treatment algorithms currently employed in the management of these patients?
- Proportion of non-operatively managed patients?
- Proportion of surgical patients approached laparoscopically?
- Recurrence rate within 6 months?

### **Secondary Research Questions**

- What is the incidence and etiology of virgin abdomen SBO?
- What is the incidence of early postoperative SBO?
- What is the success rate for non-operative management?
- What is the prevalence of complications and treatment failure in the nonoperative management of SBO?
- Proportion of patients that underwent WSOC challenge, and under what indications?
- What are the Patient Related Outcomes results?

#### Inclusion and Exclusion Criteria

#### **Inclusion Criteria:**

Adult patients (≥16 years of age) admitted for mechanical small bowel obstruction. Example etiologies which should be included:

Adhesions.

Hernias with bowel compromise (incisional/parastomal, ventral, inguinal, femoral, obturator, internal).

Malignancy (primary: lymphoma, carcinoid, GIST, adenocarcinoma/metastatic disease: colon, ovarian, gastric, pancreatic, melanoma and others).

Enteroliths/gallstones/bezoars/foreign bodies

Radiation.

Inflammation (Crohn's disease, mesenteric adenitis, appendicitis, diverticulitis, tuberculosis, actinomycosis, ascariasis).

Congenital (malrotation, duplication cysts).

Trauma (hematomas, ischemic strictures).

#### Exclusion criteria:

Functional small bowel obstruction (dysmotility or adynamic ileus secondary to abdominal operations, peritonitis, trauma or medications).

#### Center eligibility

All hospitals/units performing general surgery are eligible to join this audit. No unit size or case throughput stipulations are made. Any clinical center is welcome to participate so long as the protocol is adhered to. Countries outside Europe are eparticipate in this audit.

All participating centers will be required to register their details with the ESTES cohort study office and will be responsible for their own local approvals process prior to the start of the data collection period. Inclusion of data sets will be subject to local approval from participating clinical Centers.

Centers should ensure that they have appropriate pathways and manpower to include all consecutive eligible patients during the study period and provide >95% completeness of data entry before locking of the study REDCap® database on the November 1st 2024.

#### Patient follow-up

The audit is designed so normal patient follow-up pathways can be used to obtain outcome data. No additional visits or changes to normal follow-up should be made. However, local investigators should be proactive in identifying post-diagnosis events (or lack thereof), within the limits of normal follow-up. These may include reviewing the patient notes (paper and electronic) during admission and before discharge to note in-hospital complications, reviewing hospital systems to check for reattendances or re-admissions, and reviewing post-operative radiology reports.

#### Data completion

This research is an observational and non-interventional audit that collects data along the usual course patient pathway. The Data Collection Instrument (DCI) has been designed to reflect common parameters. We envisage that participating clinical Centers will identify a team of 4-5 members; one Consultant (clinical 'lead' of the study), trainee surgeons or data administrators who will undertake the logistical roles as well as co-ordinate data entry.

DCI 2 (patient demographics), DCI 3, 4, 5 (past medical and surgical history) and DCI 8 and 10 (follow-up information) can be completed by any suitably qualified member of the local team. DCI 6 (Current episode emergency details) and F7 (Initial complementary exams) must be completed by or in direct conjunction with an admitting staff surgeon who was present, as DCI 9 (operation details) by a staff surgeon also present itself. It should ideally be completed as close to the end of surgery as feasible, to ensure data accuracy and completeness.

#### Missing data and retrospective patient entry

The online database has been designed to allow sites to securely access an individual patient's data throughout the study period. This means that any missing or erroneous data can be altered by the local investigators whilst the data collection period is ongoing. In order to maximize data completion and emphasize its importance to collaborators, participating Centers with >5% missing data in mandatory fields (i.e. less than 95% data completeness) will be excluded from the study.

The study design means that sites may retrospectively identify <u>eligible</u> patients that were missed primarily and for whom contemporaneous patient and operation data was not entered.

#### Data collection system and information governance

Data will be recorded on a dedicated, secure server running on the REDCap® web application. REDCap® allows for secure upload and storage of data, in compliance with European Union General Data Protection Regulation 2018 (GDPR) and the Health Insurance Portability and Accountability Act of 1996 (HIPAA) legislation.

Registered local investigators will have individual password-protected access to their unit's data entered on to REDCap®. During the running of the audit, only local data will be visible to individual investigators; other sites' data will not be accessible. It is the responsibility of each participating Center to ensure their own records comply with local data governance legislation, GDPR or HIPAA, as applicable.

### Local approvals

All data collected will measure current practice, with no changes made to normal treatment. As such, this study should be registered as an audit of current practice at each participating Center. It is the responsibility of the local team at each site to ensure that local audit approval (or equivalent) is completed for their Center. Participating Centers will be asked to confirm that they have gained formal approval at their site.

#### **Authorship**

Investigators from each individual site will be included as formal co-investigators in this research, and will be PubMed searchable and citable. The output from this research will be published by the steering group on behalf of a single corporate authorship – e.g "ESTES SnapSBO Group."

#### Publication of data

The report of this audit will be prepared in accordance with guidelines set by the STROBE (strengthening the reporting of observational studies in epidemiology) statement for observational studies8, (appendix C) Data will be published as a pool from all participating units. Subgroup analyses by disease, technique or outcome variables may be presented, but no hospital-level or surgeon-level data will be published whereby an individual patient, unit or surgeon could be identified. If local investigators would like a breakdown of their own unit's data for benchmarking purposes and local presentation/discussion, this can be made available after the end of the study; however, it will not be possible or permissible to de-anonymise patient data stored in REDCap®, in strict compliance with GDPR and HIPAA.

#### Data governance

The ESTES Cohort Studies Committee welcomes the use of the data for further research that benefits patients. Requests can be submitted to the ESTES Cohort Studies Committee. Data sharing is subject to ESTES approval and the appropriate safeguarding as determined by the ESTES. Any future sub-projects should also comply with our policy of a single corporate authorship e.g. "ESTES SnapSBO Group" or similar. However, authors' contributions will be highlighted in accordance with the recommendations for the conduct, reporting, editing, and publication of scholarly work in medical journals.

#### Financial arrangements

This study is undertaken voluntarily by participating institutions under the coordination of the Emergency Surgery Cohort Study Steering Committee. It is not anticipated that participating Centers would bear any costs. Similarly, no financial reimbursement will be made to units or investigators.

### Reference list

- 1. Bass GA, Kaplan LJ, Ryan ÉJ, Cao Y, Lane-Fall M, Duffy CC, et al. The snapshot audit methodology: design, implementation and analysis of prospective observational cohort studies in surgery. Eur J Trauma Emerg S. 2022;1–11.
- 2. Detz DJ, Podrat JL, Castro JCM, Lee YK, Zheng F, Purnell S, et al. Small bowel obstruction. Curr Prob Surg. 2021;58(7):100893.
- 3. Hernandez MC, Haddad NN, Cullinane DC, Yeh DD, Wydo S, Inaba K, et al. The American Association for the Surgery of Trauma Severity Grade is valid and generalizable in adhesive small bowel obstruction. *J Trauma Acute Care.* 2018;84(2):372–8.
- 4. Vercruysse G, Busch R, Dimcheff D, Al-Hawary M, Saad R, Seagull FJ, et al. Evaluation and Management of Mechanical Small Bowel Obstruction in Adults. [internet] *Ann Arbor (MI): Michigan Medicine University of Michigan; 2021 Apr. PMID: 34314126.*
- 5. Broek RPG ten, Krielen P, Saverio SD, Coccolini F, Biffl WL, Ansaloni L, et al. Bologna guidelines for diagnosis and management of adhesive small bowel obstruction (ASBO): 2017 update of the evidence-based guidelines from the world society of emergency surgery ASBO working group. *World J Emerg Surg.* 2018;13(1):24.
- 6. Amara Y, Leppaniemi A, Catena F, Ansaloni L, Sugrue M, Fraga GP, et al. Diagnosis and management of small bowel obstruction in virgin abdomen: a WSES position paper. *World J Emerg Surg.* 2021;16(1):36.
- 7. Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. *Annals of Surgery. 2004 Aug 1;240(2):205–13*.
- 8. Vandenbroucke JP, Elm E von, Altman DG, Gøtzsche PC, Mulrow CD, Pocock SJ, et al. Strengthening the Reporting of Observational Studies in Epidemiology (STROBE): Explanation and elaboration. *Int J Surg. 2014; 12(12): 1500–24*.
- 9. Mellor K, Hind D, Lee MJ. A systematic review of outcomes reported in small bowel obstruction research. *J Surg Res. 2018; 229: 41–50*.

# **REDCap® Data Collection Instruments**

## Data Collection Instrument 1 - Patient and Centre Demographics

| Hospital Details* | Data | Values |
|--------------------------------------------|---------|-----------------|
| Primary, Secondary or Tertiary Hospital | List | List |
| Number of Beds | Integer | 0 – 3000 |
| Number or UCI beds | Integer | 0 – 3000 |
| Emergency Theatre | List | Tick Applicable |
| Acute Surgical Assessment Unit | Binary | Yes/No |
| Number of General Surgery Consultants | Integer | 1-20 |
| Split on call (Upper + Lower GI available) | Binary | Yes/No |
| Acute Care Surgery | Binary | Yes/No |
| Is ERAS practiced in General Surgery? | Binary | Yes/No |

<sup>\*</sup>will be filled once for each center

## Data Collection Instrument 2 - Patient demographics

| Demographics | Key Name | Data Type | Values |
|---|---|---|---|
| Country Code | СС | List | List of included countries (chain, number) |
| Center ID | CID | List | List of study centers (chain, number) |
| Patient ID | PID | Chain | Country code-Centre ID-patient number (chain, number) |
| Age (years) | AGE | Integer | Number |
| Sex | SEX | List | Male, Female |
| Body Mass Index | ВМІ | Integer | Weight (Kg) Height (Cm) BMI (integer) |
| Date of Admission | DOA | Date; time | Date of index admission dd/mm/yy hh:mm |
| Date of Discharge | DOD | Date | Date of discharge from hospital |
| Length of Stay | LOS | Integer | Number of Days (Integer; calculated from the admission and discharge date) |
| Cathegory | CAT | List | Ethiology (Adhesions, Bezoar, Gallstone ileus, Hernia (primary/internal/incisional/parastomal), Stenosis (anastomotic, inflammatory/endometriosis), Tumor (primary/carcinomatosis/Radiotherapy), congenital (malrotation) |

## Data Collection Instrument 3 - Patient past medical history

| Past Medical history | Key Name | Data Type | Values |
|---|---|---|---|
| Morbid Obesity (BMI>35) | МО | Binary | Yes/No. MO if BMI > 35 |
| Diabetes Mellitus | DM | Binary | Yes/No |
| Cerebro-Vascular Disease | CVD | Binary | Yes/No |
| Chronic Obstructive Pulmonary Disease | COPD | Binary | Yes/No |
| Anticogulant/aggregant Medications | ACAM | Binary | Yes/No |
| Ischemic Heart Disease | IHD | Binary | Yes/No |
| Hypertension | НВР | Binary | Yes/No. HBP if sBP>140 or dBP >90 |
| Liver Disease | LD | Binary | Yes/No |
| Chronic Kidney Disease | CKD | Binary | Yes/No. eGFR ≤59 |
| Inmunosupression/Oral Corticosteroids/<br>Chemotherapy | CIS | Binary | Yes/No (on admission) |
| Radiotherapy | RTP | Binary | Yes/No |
| Endometriosis | END | Binary | Yes/No |
| Crohn's disease | CHRD | Binary | Yes/No |
| Abdominal malignancy | AM | Binary | Yes/No. Including Gynecologic origin |
| Abdominal malignancy origin | AMO | List | Colorectal/Gynecologic/Gastroesophageal/Hepatobiliary/Splenic/<br>Pancreatic/Urologic/Haematologic |

## Data Collection Instrument 4 - Patient past surgical history

| Past Surgical history | Key Name | Data Type | Values |
|---|---|---|---|
| Previous abdominal surgery | PAS | Binary | Yes/No (excludes abdominoplasty and cesarean section) |
| Number of previous abdominal surgeries | NPS | Integer | Number (includes gyne and hernia surgeries) |
| Appendectomy | APP | Binary | Yes/No |
| Hernia surgery | HES | Binary | Yes/No |
| SBO surgery | SBOS | Binary | Yes/No |
| Previous peritonitis | PP | Binary | Yes/No |
| Date First Surgery (if one also the last) | DFS | Date | dd/mm/yy |
| First Surgery Technique | FST | Chain | Surgical technique |
| First Surgery Category | FSC | List | Predefined: CRS, GIS, HBPS, AWS, GIN, URO, VAS, AA (appendectomy) |
| First Surgery Laparoscopy | FSL | Binary | Yes/No (including conversion) |
| First Surgery Emergency | FSE | Binary | Yes/No |
| Date Last Surgery | DLS | Date | dd/mm/yy, Only in case >1 abdominal surgery |
| Last Surgery Technique | LST | Chain | Surgical Technique |
| Last Surgery Emergency | LSE | Binary | Yes/No |
| Last Surgery Laparoscopy | LSL | Binary | Yes/No (including conversion) |
| Time Last Surgery to Episode | TLSE | Calc | DOA (dd/mm/aa) - DLS (dd/mm/aa) = in Years |

# Data Collection Instrument 5 - Patient past SBO history

| Past SBO history | Key Name | Data Type | Values |
|---|---|---|---|
| Previous SBO | PSBO | Binary | Yes/No |
| Number SBO Previous Episodes | NOE | Integer | Number |
| Date Last Episode | DLE | Date | dd/mm/yy |
| Previous WSOC challenge | PG | Binary | Yes/No |
| Previous Success Non-operative Treatment | PSCT | Binary | Yes/No |
| Previous Single Band Addesion | PSBA | Binary | Yes/No |
| Previous Small Bowel Resection | PSBR | Binary | Yes/No |
| Previous SBO Etiology | PSBOE | Chain | Previous SBO cause (Adhesions/Primary Hernia/Incisional Hernia/Parastomal Hernia/Bezoar/Radiation enteritis/Primary tumor |

## Data Collection Instrument 6 - Current episode Symptoms and signs

| Current Episode Clinical Symptoms | Key Name | Data Type | Values |
|---|---|---|---|
| Date Symptoms Start | DSS | Date; time | dd/mm/yy hh:mm |
| Abdominal Pain | SAP | Binary | Yes/No |
| Nausea | NAU | Binary | Yes/No |
| Vomiting | SV | Binary | Yes/No |
| Decreased Appetite | DAP | Binary | Yes/No |
| Constipation | SNPS | Binary | Yes/No (No pass stools) |
| Obstipation | SNPG | Binary | Yes/No (No pass gas) |
| Diarrhea | DIAR | Binary | Yes/No |
| Abdominal Distension | ADI | List | No/Mild/Severe |
| Peristalsis | SPE | List | Absent; Normal; Increased |
| Temperature | ST | Decimal | Number (ºC) i.e 36.5 |
| Heart rate | SHR | Integer | Number |
| O2 Saturation | SO2 | Integer | Number |
| Systolic Blood Pressure | SBP | Integer | Number |
| Respiratory rate | SRR | Integer | Number |
| SIRS Score | SIRS | Integer | Number (1-4) (temperature >38°C or <35°C, heart rate >90 beats/min, respiratory rate >20 breaths/min or PCO $_2$ < 32 mmHg, and WBC > 12000 cells/mm3 or <4000 cells/mm |
| SBO Type | SBOT | Binary | Complete/Incomplete (if SNPS or SNPG are Yes) |

## Data Collection Instrument 7 - Initial Complementary Exams

| Current Episode Initial Complementary Exams | Key Name | Data Type | Values |
|---|---|---|---|
| White Blood Cell Count | WBC | Integer | Number x10³ |
| Hemoglobin | НВ | Decimal | Number (g/dL) |
| Potassium | К | Decimal | Number (mEq/L) |
| Creatinine | CRE | Decimal | Number (mg/dL) |
| CRP | CRP | Decimal | Number (mg/L) |
| INR | INR | Decimal | Number (mg/L) |
| Lactate | LAC | Decimal | Number (mg/dL) |
| Date First Plain Abdominal X ray | DFXR | Date; time | dd/mm/yy hh:mm |
| First AXr Stand up | FXRS | Binary | Yes/No |
| First AXr Air-Fluid Levels | FXRAF | Binary | Yes/No |
| First AXr Gastric Distension | FXRGD | Binary | Yes/No |
| First AXr Colonic Gas | FXRCG | Binary | Yes/No |
| Date Computed Tomography | DCT | Date; time | dd/mm/yy hh:mm |
| Computed Tomography Type | CTT | List | None; Without Contrast; IV Contrast; Oral Contrast; Double Contrast |
| CT Report Free Fluid | CTFF | Binary | Yes/No |
| CT Report Disminished Bowel Enhancement | CTDBE | Binary | Yes/No |
| CT Report Pneumatosis | СТР | Binary | Yes/No |
| CT Report Portal Gas | CTPG | Binary | Yes/No |
| CT Report Pneumoperitoneum | CTN | Binary | Yes/No |
| CT Report Small Bowel Wall Thickness | CTBWT | Decimal | Number (milimeters) |
| CT Report Small Bowel Diameter | CTSBD | Decimal | Number (Centimeters) |
| CT Report Feces Sign | CTFS | Binary | Yes/No (breadcrumb sign) |
| CT Report Peak Sign | CTPS | Binary | Yes/No (visible caliber change) |
| CT Report Whirl Sign | CTWS | Binary | Yes/No |
| CT Report Etiological Diagnosis | CTED | Binary | Yes/No (reported) |
| CT Report Diagnosis | CTE | Chain | Diagnosis (ie: single adhesion, matted adhesions, Hernia, Tumor) |
| AAST SBO | AAST | List | I, II, III, IV, V |

## Data Collection Instrument 8 - Current episode, course evolution

| Current Episode Course Evolution | Key Name | Data Type | Values |
|---|---|---|---|
| Severity Signs | CESS | Binary | Yes/No (if one is present: Unstable hemodynamics, peritonitis, sepsis (SIRS>2), acidosis, high lactate) |
| Ischemia Radiologic Signs | IRS | Binary | Yes/No (if one is YES: CTFF, CTDBE, CTP, CTPG, CTN, CTBWD>3mm, mesenteric edema) |
| Nasogastric/nasojejunal tube Insertion | NGTI | Binary | Yes/No |
| Initial NGT debit | INGTD | Integer | Number (mL) |
| Antibiotic Prophylaxis | PXATB | Binary | Yes/No |
| Antibiotic Treatment (if > 1 day) | TTATB | Binary | Yes/No |
| Treatment Fluids (ml/first 24h) | TTFL | Decimal | Number (ºC) |
| Treatmet Steroids | TTST | Binary | Yes/No |
| Total Urinary Output | TUO | Decimal | Number |
| WSOC Challenge | GGF | Binary | Yes/No |
| Exclusion Criteria for WSOC | GGFEC | List | No/Pregnancy/Inflamatory Bowel disease/Incarcerated hernia/Previous<br>Radiotherapy/Mechanic inflammatory ileus/Tumor or carcinomatosis/Early<br>postoperative period<1month/allergy to GGF) |
| Date WSOC | GGFD | Date; time | dd/mm/yy hh:mm |
| Post WSOC Vomiting | GGFPV | Binary | Yes/No |
| Post WSOC NGT debit | GGFNG | Decimal | Number (ºC) |
| Total Number of simple Abdominal X Ray | NXR | Integer | Number |
| Date Last Simple Abdominal X Ray | DLXR | Date; time | dd/mm/yy hh:mm |
| Last AX Ray WSOC in Stomach | LXR GGFS | Binary | Yes/No |
| Last AX Ray Deterioration | LXRD | Binary | Yes/No |
| Last AX Ray Colonic Air | LXRCA | Binary | Yes/No |
| Last AX Ray Colonic WSOC | LXRGGFC | Binary | Yes/No |
| Gas Pass | GP | Binary | Yes/No |
| Date Gas Pass | DGP | Date; time | dd/mm/yy hh:mm |
| Stools Pass | SP | Binary | Yes/No |
| Date Pass Stools | DSP | Date; time | dd/mm/yy hh:mm |
| Date Start Oral Feeding | DSOF | Date; time | dd/mm/yy hh:mm |
| Date Discharge from Emergency | DDE | Date; time | dd/mm/yy hh:mm |
| Emergency Department Lenght of Stay | EDLOS | Integer | Hours (calculation DDE-DOA) |
| Non-operative Treatment Success | COTS | Binary | Yes/No |

## Data Collection Instrument 9 - Current episode Surgery

| Current Episode Surgery | Key Name | Data Type | Values |
|---|---|---|---|
| Surgery Indicated Without Non-operative Attempt | SIWA | Binary | Yes/No |
| Date of Surgery | DSU | Date; time | dd/mm/yy hh:mm |
| Time to Surgery | TTSU | Integer | Hours (calculation DSU-DOA) |
| Laparoscopy | LAP | Binary | Yes/No (initiated) |
| Conversion | LAPC | Binary | Yes/No |
| Operative Time | ОТ | Integer | Number (Minutes) |
| Single Band Adhesilysis | SBA | Binary | Yes/No |
| Peritoneal Adhesion Index | PAI | Integer | Number |
| Ischemic Bowel | IB | Binary | Yes/No |
| Perforated Bowel | РВ | Binary | Yes/No |
| Serosal Tear | SUST | Binary | Yes/No (if one at least) |
| Unintended Bowel Perforation | UBP | Binary | Yes/No (if handmade) |
| Bowel Resection | SUBR | Binary | Yes/No |
| Anastomosis | SUBA | Binary | Yes/No |
| Stoma | SUST | Binary | Yes/No |
| Damage control (Open Abdomen) | SUDC | Binary | Yes/No |
| Hernia Repair | SUHR | Binary | Yes/No |

## Data Collection Instrument 10 - Current episode, Final outcome

| Current Episode Outcome | Key Name | Data Type | Values |
|---|---|---|---|
| Postoperative Complication | РОСО | Binary | Yes/No (if one at least) |
| Broncoaspirative pneumonia | BAP | Binary | Yes/No |
| New Acute Kidney Insufficiency | NAKI | Binary | Yes/No |
| New Onset Cardiac Arrhythmia | NOCA | Binary | Yes/No |
| Deep Vein Thrombosis/Pulmonary Embolism | DVT | Binary | Yes/No |
| Superficial Surgical Site Infection | SSSI | Binary | Yes/No |
| Deep Surgical Site Infection | DSSI | Binary | Yes/No |
| Organ Space Surgical Site Infection | OSSSI | Binary | Yes/No |
| Anastomotic leak | AL | Binary | Yes/No |
| Reoperation | RELAP | Binary | Yes/No |
| Most Severe Complication | MSCO | Chain | Named |
| Clavien Dindo | CLDI | List | I, II, IIIa, IIIb, IVa, IVb, V |
| ICU | ICU | Binary | Yes/No |
| ICU Date of Admission | ICUDOA | Date; time | Date of ICU admission dd/mm/yy hh:mm |
| ICU Date of Discharge | ICUDOD | Date; time | Date of discharge from ICU dd/mm/yy h:mm |
| ICU Lenght of Stay | ICULOS | Integer | ${\it Number of Days (Integer; calculated from the admission and discharge date)}$ |
| Death | RIP | Binary | Yes/No |
| Readmission during study period | READ | Binary | Yes/No (if after episode) |